CLINICAL TRIAL: NCT01936558
Title: The Origin of Phantom Limb Sensation and Phantom Limb Pain in Amputees
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201210078RIC
Record Dates: First submitted 2013-05-01; First posted 2013-09-06 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Exposure to Infrared Radiation

STUDY DESIGN:
Observational Model: Case-Control
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Amputees: Amputee with one arm or one leg amputated/ Far infrared ray to the phantom limb site
  Interventions: Other: Far infrared ray to the sole
- Healthy subjects: Healthy subjects under 30 years old/ Far infrared ray to the sole
  Interventions: Other: Far infrared ray to the sole

INTERVENTIONS:
Other: Far infrared ray to the sole — exposure 40-minute far infrared ray to the sole for each person/amputee.

SUMMARY:
With the far infrared ray applied to the 'phantom limbs' in amputees and the corresponding normal legs in healthy subjects, the sensation of (phantom) limb will be assessed for each subject using the techniques of fMRI and meridian response.

DETAILED DESCRIPTION:
This project will investigate two main hypotheses based on our previous studies on phantom limb sensation and phantom limb pain. The first hypothesis states that phantom limb sensation and phantom limb pain both correlate with the 'phantom limb', while the second one maintains that the phantom limb can interact with the patient's body by means of the meridian system. With the far infrared ray applied to the 'phantom limbs' in amputees and the corresponding normal legs in healthy subjects, the sensation of (phantom) limb will be assessed for each subject using the techniques of fMRI and meridian response. By analyzing the data collected from both groups, the investigators expect both hypotheses will be supported by the results of experiments in this project.

ELIGIBILITY:
Inclusion Criteria:

* Amputees: at least one arm or one leg amputated
* Healthy subjects: healthy person under 30 years old

Exclusion Criteria:

* with mental diseases

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Amputees / healthy subjects
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Resting functional MR images | one year
  The resting fMRI images will be obtained before and after the far infrared exposed to the phantom limb site. The default mode of the brain will be analyzed. If the default mode was changed, it was one of the evidence that the neural signal was transmitted from the phantom limb site into the brain and caused the change.

CONTACTS AND LOCATIONS:
Overall Officials: Rong-Sen Yang, Study Chair — Department of orthopedics, NTUH
Locations (1):
- NTUH department of orthopedics; NTU department of electrical engneering, Taipei, Taiwan, Taiwan